CLINICAL TRIAL: NCT05342740
Title: A Multicenter Case Control Study of Biomarkers in Diabetic Chronic Wounds Based on Combined Multi-omics Analysis Techniques
Brief Title: Study of Biomarkers in Diabetic Chronic Wounds
Status: Recruiting | Type: Observational
Sponsor: Yibing Wang (Other)
Responsible Party: Sponsor-Investigator, Yibing Wang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(013)
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Biomarker; Chronic Wound
Keywords: chronic diabetic wound; early diagnosis; prognostic; prediction; biomarker; muti-omics
MeSH Terms: conditions — Diabetes Mellitus; Disease | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group-CWD: diabetic patients with chronic wounds (CWD)
  Interventions: Other: collect whole blood, urine and stool samples
- Control group 1-ND: patients without diabetes (ND)
  Interventions: Other: collect whole blood, urine and stool samples
- Control group 2-NWD: diabetic patients without newly identified wound (NWD)
  Interventions: Other: collect whole blood, urine and stool samples

INTERVENTIONS:
Other: collect whole blood, urine and stool samples — collect whole blood, urine and stool samples

SUMMARY:
This study aims to discover, verify and evaluate the potential biomarkers with regard to the diagnosis, prognostic and/or prediction of diabetic chronic wounds.

DETAILED DESCRIPTION:
Investigators will conduct a multicenter prospective case control study consisting of three stages.

In the first stage, investigators will collect clinical data and blood, urine and stool samples from diabetic patients with chronic wound (CWD), diabetic patient without newly identified wound (NWD) and patients without diabetes (ND to discover the candidate bioindicator with differences through combined high-throughput non targeted detection.

In the second stage, investigators will expand the sample size and collect the clinical data and biological samples (blood, urine and stool) of the CWD,NWD and ND participants to verify the difference of the candidate bioindicator in the first stage by targeted technologies.

In the third stage, investigators will collect the clinical data and biological samples (blood, urine and stool) of the CWD and NWD participants to evaluate the value of these candidate bioindicators as biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75;
2. Signed the informed consent form；
3. Subjects in the ND group are the healthy participants without diabetes；
4. Subjects in the NWD group are the diabetic participants without newly identified wounds；
5. Subjects in the CWD group are the diabetic participants with chronic wounds

Exclusion Criteria:

1. With sever acute underlying diseases of the brain, heart, lungs, liver and/or kidney;
2. No diabetes but combined with lower limb arterial stenosis, occlusion or other conditions affecting wound healing or other causes of wounds such as varicose veins in the lower limbs;
3. Special exclusion criteria for blood, urine and stool samples taking.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are required to complete a structured questionnaire for assessment of inclusion requirement and then divided into the CWD group, NWD group and the ND group.
Sampling Method: Probability Sample
Enrollment: 930 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bioindicators with differences among groups | Through study completion, an average of 1 year
  Analysis omics results and discover candidate bioindicators that differ between groups
Basic clinical and demographic information of participants in groups | Through study completion, an average of 1 year
  Collect basic clinical and demographic information of participants in groups by a CRF

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yibing, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No